CLINICAL TRIAL: NCT04853043
Title: APK Mutant: A Single Arm Phase II Study of Cetuximab in Third Line for Mutant APC, TP53 and RAS Patients With Refractory Metastatic Colorectal Cancer
Brief Title: Cetuximab in Third Line for Mutant APC, TP53 and RAS Patients With Refractory Metastatic Colorectal Cancer
Acronym: APK Mutant
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI Determination - Slow recruitment, funding concerns, poor response to treatment
Sponsor: University of Utah (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI141689; R21CA252436 (NIH)
Record Dates: First submitted 2021-04-16; First posted 2021-04-21 (Actual); Results first posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Intervention Model Description: Single arm, open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cetuximab (Experimental)
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Drug: Cetuximab — Cetuximab will be administered every 2 weeks (14 days). The initial dose of 500 mg/m2 is to be administered by IV infusion over 120 minutes on the first day of the treatment. In the absence of infusion reactions, subsequent doses are to be administered over 60 minutes biweekly. Each cycle will be defined as 14 days of treatment.

SUMMARY:
A prospective, multi-center, phase II study of 21 patients to evaluate the efficacy of the epidermal growth factor receptor (EGFR) inhibitor, Cetuximab in patients with metastatic colorectal cancer (mCRC) harboring Adenomatous polyposis coli (APC), tumor protein p53 (TP53) and RAS mutations.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged ≥ 18 years.
* Histologically confirmed metastatic colorectal adenocarcinoma with mutant APC, TP53 and KRAS genes as determined by the local Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory are eligible. All RAS mutations are allowed (KRAS, Neuroblastoma RAS (NRAS), HRAS). Patients with wild type KRAS, APC or TP53 are ineligible.
* Progression or unwanted toxicities on at least 2 prior lines of treatment including 5-Fluorouracil, oxaliplatin and irinotecan-based regimen
* Study participants must have measurable disease by RECIST 1.1 criteria by CT or MRI.
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2.
* Study participants with treated and/or stable brain metastases are allowed
* Study participants must have anticipated life expectancy > 3 months
* Adequate organ function as defined as:

  * Hematologic:

    * Absolute neutrophil count (ANC) ≥ ≥1000/µL
    * Platelet count ≥ 100,000/mm3
    * Hemoglobin ≥ 9 g/dL
  * Hepatic:

    * Serum Bilirubin ≤ 2 x ULN or ≤ 3 x ULN for subjects with Gilbert's syndrome
    * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3.0 times the upper limit of normal (ULN; or 5.0 times the ULN in the setting of liver metastases)
  * Renal:

    * Serum creatinine ≤1.5 times the ULN, or creatinine clearance (measured via 24-hour urine collection) ≥40 mL/minute (that is, if serum creatinine is >1.5 times the ULN, a 24-hour urine collection to calculate creatinine clearance must be performed)
* For female subjects: Negative pregnancy test or evidence of post-menopausal status. The post-menopausal status will be defined as having been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women < 50 years of age:

    * Amenorrheic for ≥ 12 months following cessation of exogenous hormonal treatments; and
    * Luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution; or
    * Underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
  * Women ≥ 50 years of age:

    * Amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments; or
    * Had radiation-induced menopause with last menses >1 year ago; or
    * Had chemotherapy-induced menopause with last menses >1 year ago; or
    * Underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy).
* Female subjects of childbearing potential and male subjects with a sexual partner of childbearing potential must agree to use a highly effective method of contraception throughout the study and for at least 12 months after last study treatment administration.
* Male subjects must agree to use a condom during intercourse for the duration of study therapy and for at least 12 months after last study treatment administration.
* Recovery to baseline or ≤ Grade 1 CTCAE v5.0 from toxicities related to any prior cancer therapy, unless considered clinically not significant by the treating investigator.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* Prior use of systemic anti-EGFR therapy including cetuximab or panitumumab is not allowed but prior use irinotecan, oxaliplatin, regorafenib or Trifluridine/Tipiracil (TAS-102) is allowed
* Study participants with prior or concurrent malignancy whose natural history or treatment have the potential to interfere with the safety or efficacy assessment of the investigational regimen, as determined by the investigator
* Study participants with new or progressive brain metastases (active brain metastases) or leptomeningeal disease who need immediate central nervous system (CNS)-specific treatment during first cycle of treatment as determined by the treating physician.

  --Note: Brain metastases or cranial epidural disease adequately treated with radiotherapy and/or surgery and stable for at least 4 weeks before the first dose of study treatment will be allowed on trial. Subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of the first dose of study treatment.
* Current evidence of uncontrolled, significant intercurrent illness including, but not limited to, the following conditions:

  * The patient has clinically relevant coronary artery disease or history of myocardial infarction in the last 12 months or high risk of uncontrolled arrhythmia or uncontrolled cardiac insufficiency.
  * The patient has uncontrolled or poorly-controlled hypertension (>180 mmHg systolic or > 130 mmHg diastolic.
  * Any other condition that would, in the Investigator's judgment, contraindicate the subject's participation in the clinical study due to safety concerns or compliance with clinical study procedures (e.g., infection/inflammation, intestinal obstruction, unable to swallow medication, [subjects may not receive the drug through a feeding tube], social/ psychological issues, etc.)
* Known HIV infection with a detectable viral load within 6 months of the anticipated start of treatment.

  --Note: Subjects on effective antiretroviral therapy with an undetectable viral load within 6 months of the anticipated start of treatment are eligible for this trial.
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination, radiographic findings, and tuberculosis (TB) testing in line with local practice), hepatitis B (known positive hepatitis B virus (HBV) surface antigen (HBsAg) result), or hepatitis C.

  --Note: Subjects with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody (anti-HBc) and absence of HBsAg) are eligible. Subjects positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Medical, psychiatric, cognitive, or other conditions that may compromise the subject's ability to understand the subject information, give informed consent, comply with the study protocol or complete the study.
* Known prior severe hypersensitivity attributed to compounds of chemical or biologic composition similar to those of cetuximab, or if the patient had red meat allergy/tick bite history (NCI CTCAE v5.0 Grade ≥ 3).
* Live attenuated and inactive vaccinations within 4 weeks of the first dose of study treatment and while on trial is prohibited. Coronavirus Disease 19 (COVID-19) vaccines are allowed
* The patient is pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vaia Florou, MD, Principal Investigator — Huntsman Cancer Institute
Locations (2):
- United States (2):
  - Intermountain Medical Center, Salt Lake City, Utah
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cetuximab
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cetuximab
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.71 (8.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7
Eastern Cooperative Oncology Group (ECOG) [Count of Participants; unit: Participants]
  0 Fully active | 0
  1 Restricted | 7
  2 Ambulatory | 0
  3 Limited selfcare | 0
  4 Completely disabled | 0
  5 Dead | 0
Height [Mean (Standard Deviation); unit: cm] | 167.13 (10.17)
Weight [Mean (Standard Deviation); unit: kg] | 88.34 (33.94)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.02 (10.25)

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Evaluate the PFS among patients treated with cetuximab in APC, TP53 and RAS mutated refractory metastatic colorectal cancer.
  PFS will be measured from the date of first dose of study drug until the first documented radiographic evidence of disease progression by Response Evaluation Criteria In Solid Tumors Criteria (RECIST) criteria 1.1, clinical progression per investigator judgement, start of new anti-cancer therapy, or death from any cause.
  Per RECIST 1.1 for target lesions, Progressive Disease (PD) is a >=20% increase in the sum of the longest diameter (LD) of target lesions.
  Disease progression by RECIST 1.1 is PD.
Time Frame: PFS will be measured from the date of first dose of study drug until first documented clinical or radiographic evidence of disease progression by RECIST 1.1, clinical progression, start of new therapy or death. Estimated assessment at 6 months.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Cetuximab
Number analyzed (Participants) | 7
days | 48 [27.68 to 54.04]

2. Secondary Outcome: Overall Survival (OS).
Description: Evaluate the overall survival (OS) among patients treated with cetuximab in APC, TP53 and RAS mutated refractory metastatic colorectal cancer.
  Upon discontinuation of study therapy, subjects will be followed for survival from the date of study therapy initiation until death, end of the study, or subject withdrawal of consent, whichever comes first.
Time Frame: OS was measured from the date of first dose of study drug until death from any cause (up to 223 days)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Cetuximab
Number analyzed (Participants) | 7
days | 94.50 [54.74 to 158.26]

ADVERSE EVENTS:
Time Frame: Adverse events were followed until 30 days (± 7 days) after the last dose of study drug (up to 112 days after initiation of study treatment). Survival was followed from the date of the first dose of study drug until death from any cause (up to 223 days after initiation of study treatment).
Arm/Group | Cetuximab
All-Cause Mortality (participants affected / at risk) | 7/7
Serious Adverse Events (participants affected / at risk) | 3/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetuximab (N=7)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Alkaline phosphatase increased (Gastrointestinal disorders) | 2 (2)
Colonic obstruction (Gastrointestinal disorders) | 2 (2)
Electrocardiogram QT corrected interval prolonged (Gastrointestinal disorders) | 2 (2)
Hypokalemia (Nervous system disorders) | 2 (2)
Small intestinal obstruction (Metabolism and nutrition disorders) | 3 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetuximab (N=7)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Alanine aminotransferase increased (Gastrointestinal disorders) | 1 (1)
Alkaline phosphatase increased (Gastrointestinal disorders) | 1 (1)
Anemia (Gastrointestinal disorders) | 2 (2)
Anorexia (Gastrointestinal disorders) | 3 (5)
Ascites (Gastrointestinal disorders) | 3 (3)
Aspartate aminotransferase increased (Gastrointestinal disorders) | 1 (1)
Back pain (Gastrointestinal disorders) | 1 (1)
Blood and lymphatic system disorders - Other, specify (Gastrointestinal disorders) | 1 (1)
Blood bicarbonate decreased (Gastrointestinal disorders) | 1 (1)
Blood bilirubin increased (Gastrointestinal disorders) | 2 (2)
Bullous dermatitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Creatinine increased (Gastrointestinal disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Disease progression (Gastrointestinal disorders) | 2 (2)
Edema limbs (Gastrointestinal disorders) | 1 (1)
Encephalopathy (Gastrointestinal disorders) | 1 (1)
Fatigue (Gastrointestinal disorders) | 3 (3)
Fever (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 5 (5)
Hematuria (Nervous system disorders) | 2 (2)
Hepatobiliary disorders - Other, specify (Nervous system disorders) | 1 (1)
Hot flashes (Nervous system disorders) | 1 (1)
Hypercalcemia (Nervous system disorders) | 1 (1)
Hyperglycemia (Nervous system disorders) | 1 (1)
Hyperkalemia (Nervous system disorders) | 1 (1)
Hypoalbuminemia (Nervous system disorders) | 2 (2)
Hypocalcemia (Nervous system disorders) | 1 (1)
Hypokalemia (Nervous system disorders) | 1 (2)
Hyponatremia (Nervous system disorders) | 2 (2)
Infusion related reaction (Nervous system disorders) | 1 (1)
Insomnia (Nervous system disorders) | 3 (4)
Leukocytosis (Nervous system disorders) | 1 (1)
Lipase increased (Nervous system disorders) | 1 (1)
Lymphocyte count decreased (Nervous system disorders) | 1 (1)
Metabolism and nutrition disorders - Other, specify (Nervous system disorders) | 1 (1)
Nail changes (Nervous system disorders) | 1 (1)
Nausea (Nervous system disorders) | 2 (3)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1)
Pain (Nervous system disorders) | 1 (1)
Pain in extremity (Nervous system disorders) | 1 (1)
Proteinuria (Nervous system disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 (6)
Rash maculo-papular (Metabolism and nutrition disorders) | 2 (2)
Respiratory, thoracic and mediastinal disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1)
Sepsis (Metabolism and nutrition disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (2)
Skin and subcutaneous tissue disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1)
Small intestinal obstruction (Metabolism and nutrition disorders) | 1 (1)
Surgical and medical procedures - Other, specify (Metabolism and nutrition disorders) | 1 (1)
Vaginal hemorrhage (Metabolism and nutrition disorders) | 1 (1)
Vomiting (Metabolism and nutrition disorders) | 3 (3)
Weight loss (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Each party shall have the right to publish and disseminate information derived from the performance of the Statement of Work.

Qualification for authorship shall be in keeping with generally accepted criteria. Intermountain Health Services shall provide the University of Utah with a copy of any proposed publication for review and comment at least thirty (30) days prior to submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/43/NCT04853043/Prot_SAP_000.pdf